CLINICAL TRIAL: NCT03307720
Title: Agonist Trigger Versus Classical HCG Trigger in Controlled Ovarian Stimulation Among Three Different Subsets of Patients (Poor Responders, Normoresponders and High Responders)
Brief Title: Agonist Versus Classical HCG Trigger (Poor Responders, Normoresponders and High Responders)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ginegorama S.L. (Other)
Responsible Party: Principal Investigator, Gorka Barrenetxea, Professor of Gynecology & Obstetrics Universidad del País Vasco/Euskal Herriko Unibertsitatea. Medical Director of Reproducción Bilbao, Ginegorama S.L.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGONIST TRIGGER
Record Dates: First submitted 2017-09-30; First posted 2017-10-12 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Ovulation Induction; In Vitro Fertilization (IVF); Infertility, Female; Oocytes
Keywords: agonist trigger; Ovulation induction; Controlled ovarian stimulation (COS); Poor responder
MeSH Terms: conditions — Infertility, Female | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Intervention Model Description: IVF patients enrolled either to HCG or agonist trigger ovulation induction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Poor responders. Classical trigger (Active Comparator): Intervention: HCG trigger (Administration of recombinant HCG 250 UI subcutaneously 36 prior to oocyte retrieval.
  Women scheduled for IVF treatment with 4 or less antral follicles in ultrasound assessment.
  Interventions: Drug: Human chorionic gonadotropin
- Poor responders. Agonist trigger (Experimental): Intervention: Agonist trigger (administration of 0,2 mg of Triptoreline subcutaneously 36 hours prior to oocyte retrieval)
  Women scheduled for IVF treatment with 4 or less antral follicles in ultrasound assessment.
  Interventions: Drug: Gonadotropin Releasing Hormone Agonists (GNRH-A)
- Normo responders. Classical trigger (Active Comparator): Intervention: HCG trigger (Administration of recombinant HCG 250 UI subcutaneously 36 prior to oocyte retrieval.
  Women scheduled for IVF treatment with more than 4 and less than 16 antral follicles in ultrasound assessment.
  Interventions: Drug: Human chorionic gonadotropin
- Normo responders. Agonist trigger (Experimental): Intervention: Agonist trigger (administration of 0,2 mg of Triptoreline subcutaneously 36 hours prior to oocyte retrieval)
  Women scheduled for IVF treatment with more than 4 and less than 16 antral follicles in ultrasound assessment.
  Interventions: Drug: Gonadotropin Releasing Hormone Agonists (GNRH-A)
- High responders. Classical trigger (Active Comparator): Intervention: HCG trigger (Administration of recombinant HCG 250 UI subcutaneously 36 prior to oocyte retrieval.
  Women scheduled for IVF treatment with more than 15 antral follicles in ultrasound assessment.
  Interventions: Drug: Human chorionic gonadotropin
- High responders. Agonist trigger (Experimental): Intervention: Agonist trigger (administration of 0,2 mg of Triptoreline subcutaneously 36 hours prior to oocyte retrieval)
  Women scheduled for IVF treatment with more than 15 antral follicles in ultrasound assessment.
  Interventions: Drug: Gonadotropin Releasing Hormone Agonists (GNRH-A)

INTERVENTIONS:
Drug: Gonadotropin Releasing Hormone Agonists (GNRH-A) — Administration of a gonadotropin releasing hormone agonist (GnRH-a) (0,2 ml) subcutaneously, 36 hours before ovum pick-up in IVF treatments.
  Other Names: Agonist trigger
  Arms: High responders. Agonist trigger; Normo responders. Agonist trigger; Poor responders. Agonist trigger
Drug: Human chorionic gonadotropin — Administration of Human chorionic gonadotropin (HCG) 250 IU subcutaneously , 36 hours before ovum pick-up in IVF treatments.
  Other Names: HCG trigger
  Arms: High responders. Classical trigger; Normo responders. Classical trigger; Poor responders. Classical trigger

SUMMARY:
Agonist triggering in controlled ovarian stimulation protocols is being used during last years (among high responder patients to avoid OHSS).

Indeed, agonist triggering is more physiologic than HCG triggering. Investigators propose to compare the effectiveness of both types of trigger among three different subsets of patients:

1. Poor responders.
2. Normo-responders
3. High responders Comparing both the number and the quality of achieved oocytes.

DETAILED DESCRIPTION:
During the last years, ovulation triggering in controlled ovarian stimulation protocols has been used specially to avoid hyperstimulation syndromes (OHSS). Indeed, the substitution of the classical HCG triggering by the agonist one, reduces almost to zero the risk of OHSS.

On the other hand poor responder patients to ovarian stimulation represent a challenge in assisted reproduction. Defining poor responders is not easy, but we can define them as those patients with less than 4 eggs obtained after oocyte retrieval.

Different strategies have been proposed to overcome this problem. In other words, to obtain more oocytes. These include an increase in FSH doses, an increase in FSH action by adding sensitizers agents.

Among the possible strategies, investigators propose the agonist triggering. HCG (classical) triggering represents the use of a LH-like product (with a prolonged action). The administration of a GnRH agonist provoke the production and liberation of both FSH and LH. Thus, the pro-ovulatory action is more physiologic , and possibly, more effective.

So, the use of a triggering protocol that nowadays is being used among high responders (thus reducing the OHSS risk) is proposed for both poor responder and normo-responder patients trying to achieve more oocytes, and specifically more mature oocytes.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for IVF treatment.
* First ovarian stimulation
* Two ovaries present
* No previous ovarian surgery
* No contraindication for any of the assigned treatments

Exclusion Criteria:

* Previous ovarian surgery.
* Previous IVF treatments.
* Absence of one ovary
* Presence of an endometrioma

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-18 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Mature oocytes | Up to 24 weeks
  Number of mature oocytes achieved after oocyte retrieval.

SECONDARY OUTCOMES:
Relation mature oocytes/punctured oocytes | Up to 24 weeks
  Relation between the number of mature oocytes and the follicles.
Fertilized oocytes | Up to 24 weeks
  Number of fertilized oocytes
Relation fertilized oocytes/achieved Mature oocytes | Up to 24 weeks
  Relation between the number of fertilized oocytes and the mature oocytes achieved.
Number of blastocysts developed | Up to 24 weeks
  Number of blastocysts developed in each arm of the study.
Cancelled cycles | Up to 24 weeks
  Percentage of cancelled cycles

CONTACTS AND LOCATIONS:
Overall Officials: Gorka Barrenetxea, PhD, Principal Investigator — Reproducción Bilbao. Universidad del País Vasco/Euskal Herriko Unibertsitatea; Jon Iker Arambarri, MD, Study Chair — Reproducción Bilbao. Universidad del País Vasco/Euskal Herriko Unibertsitatea
Locations (1):
- Reproduccion Bilbao Assisted Reproduction Center, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No